CLINICAL TRIAL: NCT06015048
Title: A Phase 1b/2 Study to Evaluate the Safety, Tolerability and Efficacy of SHR-A1811 Combined With Other Antitumor Therapies in Advanced Solid Tumors.
Brief Title: A Trial of SHR-A1811 Combined With Other Antitumor Therapies in Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-208
Record Dates: First submitted 2023-08-01; First posted 2023-08-29 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: HER2-expressing Advanced Solid Tumors
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Intervention: Drug: SHR-A1811 combined with Pyrotinib (Experimental)
  Interventions: Drug: SHR-A1811 combined with Pyrotinib.
- Part B1: Intervention: Drug: SHR-A1811 combined with other antitumor therapies (Experimental)
  Interventions: Drug: SHR-A1811 combined with other antitumor therapies

INTERVENTIONS:
Drug: SHR-A1811 combined with Pyrotinib. — SHR-A1811 combined with Pyrotinib
  Arms: Part A: Intervention: Drug: SHR-A1811 combined with Pyrotinib
Drug: SHR-A1811 combined with other antitumor therapies — SHR-A1811 combined with other antitumor therapies
  Arms: Part B1: Intervention: Drug: SHR-A1811 combined with other antitumor therapies

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-A1811 combined with other antitumor therapies in advanced solid tumors. To explore the reasonable dosage of SHR-A1811 combined with other antitumor therapies for advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent. Have good compliance and cooperated with follow-up visits.
2. Subjects are older than or equal to 18 years old and younger than or equal to 75 years old on the day of signing the informed consent. Male or female.
3. ECOG score 0-1.
4. Life expectancy is at least 12 weeks.
5. Histologically or cytologically confirmed metastatic or advanced unresectable HER2-expression or Her-2 functional mutations solid tumors.
6. Provide ≥ 6(or ≥8)sections of formalin-fixed, paraffin-embedded tumor tissue blocks or unstained tumor specimen sections. Sections should be archived within 1 year before the first study treatment or freshly obtained (freshly obtained is preferred).
7. ≥1 Measurable lesions, according to the Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1. The dose escalation phase allows for the absence of measurable lesions.
8. Organ function met criteria within 7 days prior to initial administration (No blood component or cell growth factor was used within 14 days before the initial administration):
9. Left ventricular ejection fraction (LVEF) ≥ 50% at baseline within 28 days prior to initial administration.
10. Males and women of childbearing age must use reliable contraception from the written informed consent to 7 months after last drug administration (SHR-A1811) or 8 weeks after last drug administration (Pyrotinib) or 6 months after last drug administration (BP102 or Oxaliplatin or Calcium levonofolinate or fluorouracil), the latest time should be taken as final. Women of childbearing age must have had a pregnancy test (serum or urine) with negative results within 7 days prior to initial administration and must not in lactation period.

Exclusion Criteria:

1. Subjects with untreated or known active CNS metastasis. Subjects with a history of meningeal metastasis or known active meningeal metastasis.
2. Have a history of antibody drug conjugate with following characteristics: topoisomerase I inhibitors, including Enhertu (DS-8201a), U3-1402, etc. Part A: Have a history of Her-2 targeted tyrosine-kinase inhibitor (TKI).
3. Palliative radiotherapy within 14 days prior to initial administration. Subjects who had received systemic anti-tumor therapy within 4 weeks prior to initial administration will not permitted. The interval between the end of small-molecule targeted drugs administration and initial test drug administration must be ≥ 5 half-lives or 7 days (take the longer time). The interval between the end of Chinese patent anti-tumor drug administration and initial test drug administration must be ≥ 2 weeks. Participating in another clinical study of other drugs. The interval between the previous clinical study drug use and this study initial administration is less than 4 weeks or 5 half-lives of previous clinical study drug (take the shorter time).
4. Toxicity and/or complications of previous interventions were not recovered to NCI-CTCAE ≤ grade 1 or didn't meet this inclusion criteria and exclusion criteria. If investigator determines that the toxicity and/or complications are NCI-CTCAE ≤ grade 2 and there is no safety risk, this subject can be enrolled. For example, patients with type 1 diabetes or hypothyroidism who have been treated with immune checkpoint inhibitors and are stable after hormone replacement therapy.
5. Have a history of (non-infectious) interstitial lung disease (ILD). Suspected ILD. Other moderate and severe lung diseases that may interfere the detection or management of drug-related pulmonary toxicity and severely affect respiratory function within 3 months before the first test drug administration. Any autoimmune disease, connective tissue disease, or inflammatory disease with lung involvement.
6. Patients unable to swallow orally administered medication and other disorders likely to interfere the absorption of the study drugs within 28 days before the first test drug administration.
7. Patients with moderate and severe ascites of clinical symptoms Refractory or moderate to severe pleural effusion or pericardial effusion.
8. Patients with intestinal obstruction within 6 months prior to the first test drug administration or presence of signs and symptoms of intestinal obstruction (patients can be enrolled if surgical treatment had been performed and the obstruction had been completely resolved).
9. Have clinically significant cardiovascular disease.
10. Previous or combined with other malignancies except those have achieved complete remission and do not require or are not expected to require other treatment during the study period within at least 5 years prior to screening, including basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, cervical carcinoma in situ, local prostate cancer, ductal carcinoma in situ after radical surgery, etc (hormone therapy for non-metastatic prostate cancer or breast cancer is allowed) .
11. Serious infections within 28 days prior to the first test drug administration. Active infections that had received therapeutic intravenous antibiotics within 2 weeks prior to the first test drug administration. Prophylactic antibiotic therapy can be enrolled.
12. Active hepatitis B or active hepatitis C infection. Active hepatitis B is defined as hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥10000 copies/ml [2000 IU/ml] during screening. Active hepatitis C is defined as hepatitis C virus antibody positive and HCV-RNA positive during screening. Patients with active pulmonary tuberculosis infection within 1 year before enrolment, or with a history of active pulmonary tuberculosis infection but without regular treatment more than 1 year before enrolment. Has known immunodeficiency disorders, including human immunodeficiency virus (HIV) infection, etc. Received attenuated live vaccines within 28 days of initial administration. Expected use of attenuated live vaccines during the study period.
13. Major surgery history other than diagnostic or biopsy surgery within 28 days prior to initial administration. Minor traumatic surgery within 7 days prior to initial administration. Non-healing wounds. Untreated bone fractures.
14. Known allergy to any component of SHR-A1811. History of severe allergic reactions to other monoclonal antibody/fusion protein drugs. Part A: known allergy to any component of Pyrotinib.
15. Female subjects who are pregnant, in lactation period, or planning pregnancy during the study period.
16. Uncontrolled mental illness and other conditions which will affect the completion of the study, such as alcohol abuse, drug or substance abuse, criminal detention, etc.
17. Any other conditions that may not eligible to participate in this study according to researchers' judgment.

For Part B1, subjects must not meet any of the following supplementary criteria at the same time, otherwise they will not be enrolled in the study:

1、Presence of grade >1 peripheral neuropathy.

For those who plan to receive BP102 combination therapy, subjects must not meet any of the following supplementary criteria at the same time, otherwise they will not be enrolled in the study:

1. Bleeding tendency, coagulation dysfunction, or high risk of thrombosis.
2. Poorly controlled hypertension after medication (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg in the case of regular anti-hypertensive therapy) and prior hypertensive crisis or hypertensive encephalopathy. Severe cerebrovascular diseases and clinically significant vascular diseases.
3. Severe cerebrovascular disease, including cerebrovascular accident (CVA), transient ischemic attack (TIA), and significant vascular disease (including but not limited to aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Part A: Maximally Tolerated Dose (MTD),)(Phase ⅠB). | From the first dose to the last dose, about 11 months
Part A: recommended phase 2 dose (RP2D)(Phase ⅠB). | From the first dose to the last dose, about 11 months
Part A: Adverse Events (Phase ⅠB) | From the first dose to the last dose, about 11 months
Part A: Objective Response Rate (ORR) (Phase Ⅱ) | From the first dose to the last dose, about 11 months

SECONDARY OUTCOMES:
Part A: ORR (Phase ⅠB). | From the first dose to the last dose, about 11 months.
Part A: Disease Control Rate (DCR) (Phase ⅠB and Phase Ⅱ) | From the first dose to the last dose, about 11 months
Part A: Duration of Response (DoR) (Phase ⅠB and Phase Ⅱ) | From the first dose to the last dose, about 11 months
Part A: Progression-free survival (PFS) (Phase ⅠB and Phase Ⅱ) | From the first dose to the last dose, about 13 months.
Part A: Overall survival (OS) (Phase ⅠB and Phase Ⅱ) | From the first dose to the last dose, about 13 months
Part A: Adverse Events (PhaseⅡ). | about 11 months.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Cancer Hospital & Institute-Department of Gastrointestinal Oncology, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital-The Eighth Department of Internal Medicine, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University-Department of Medical Oncology, Zhengzhou, Henan
  - Hubei Cancer Hospital-Department of Abdominal Oncology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanxi Provincial Cancer Hospital-Gastroenterology Department, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital-Department of digestive oncology, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided